CLINICAL TRIAL: NCT02069288
Title: Effects of Fludrocortisone on Norepinephrine-mean Arterial Pressure Dose-response, Gastric Mucosal Perfusion and Arterial Stiffness in Septic Shock
Brief Title: Effects of Fludrocortisone on Norepinephrine-mean Arterial Pressure Dose-response in Septic Shock
Acronym: FLUDRO
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Problems of drugs supply by the manufacturer
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EudraCT 2007-007971-18; CIC0203/082
Record Dates: First submitted 2013-12-23; First posted 2014-02-24 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2014-02

CONDITIONS: Septic Shock
Keywords: fludrocortisone; pharmacology; septic shock
MeSH Terms: conditions — Shock, Septic | interventions — Fludrocortisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Fludrocortisone
  Interventions: Drug: Fludrocortisone
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fludrocortisone — 50 µg of fludrocortisone per os
  Other Names: 9- alpha- fluorohydrocortisone
  Arms: 1
Drug: Placebo — 1 tablet of placebo per os
  Arms: 2

SUMMARY:
Septic shock (associated with relative adrenal insufficiency) is characterized by decreased arterial responsiveness to catecholamines. The association of hydrocortisone and fludrocortisone has demonstrated an improvement in survival in septic shock patients. If hydrocortisone has shown to increase vascular responsiveness, the role of fludrocortisone remains to be elucidated. The purpose of our study is to investigate the effect of a physiological dose of fludrocortisone alone on norepinephrine-mean arterial pressure dose-response relationship, gastric mucosal perfusion and arterial stiffness in patients with septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Patients over than 18 years old
* Septic shock
* Haemodynamic stability (mean arterial pressure between 70 and 80 mmHg) for at least 1 hour, with a norepinephrine dose less than 0,5 µg/kg/min
* Written informed consent

Exclusion Criteria:

* Corticotherapy
* Known allergy to Fludrocortisone
* Esophageal or gastric disease
* Pregnant woman
* Inclusion in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Norepinephrine-mean arterial pressure dose-response relationship | 1.5 h after administration

SECONDARY OUTCOMES:
Systolic and diastolic arterial pressures, heart rate, cardiac output, systemic vascular resistances | During 3 h after administration
Central aortic pressures, Augmentation Index (Aix). | During 3 h after administration
Arterial stiffness: Carotid-femoral Pulse Wave Velocity | During 3 h after administration
Humeral diameter and distensibility | During 3 h after administration
Gastric mucosal perfusion | During 3 h after administration
Plasma electrolytes, blood glucose, serum creatinine | Each hour during 3 h after administration
Plasma renin, aldosterone, norepinephrine, epinephrine, fludrocortisone, TNF alpha concentrations | Each hour during 3 h after administration
Urinary electrolytes excretion | Each hour during 3 h after administration

CONTACTS AND LOCATIONS:
Overall Officials: Bruno LAVIOLLE, MD, Principal Investigator — Rennes University Hospital; Eric BELLISSANT, MD, PhD, Study Chair — Rennes University Hospital
Locations (1):
- Service de Réanimation Chirurgicale - Hôpital de Pontchaillou, Rennes, France